CLINICAL TRIAL: NCT00969891
Title: Population Based Pharmacokinetic and Pharmacodynamic Dosage Model for Cytarabine, Daunorubicin and Etoposide for Acute Myeloid Leukemia
Brief Title: Study of Dosage Individualisation for the Treatment of Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Mikkel Krogh-Madsen (Other)
Collaborators: Rigshospitalet, Denmark (Other); Herlev Hospital (Other)
Responsible Party: Sponsor-Investigator, Mikkel Krogh-Madsen, PhD student, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: AMLPKPD-20081127; EudraCT nummer 2008-008165-35
Record Dates: First submitted 2009-08-28; First posted 2009-09-01 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples

GROUPS / COHORTS (1):
- AML patients in induction treatment
  Interventions: Other: PK-PD analysis

INTERVENTIONS:
Other: PK-PD analysis — The danish medicines agency regards new knowledge in pharmacokinetics and pharmacodynamics as an intervention.

SUMMARY:
The present study is not hypothesis driven but will explore the ability of pharmacokinetic-pharmacodynamic modelling to predict optimal dosage of the chemotherapeutic drugs used in therapy in adult patients with acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* adult men and women with newly diagnosed acute myeloid leukemia

Exclusion Criteria:

* under age 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2009-09; Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
significant covariates from the PK study | after complete analysis of data

SECONDARY OUTCOMES:
Amount of the three drugs in patient plasma samples | within 3 months of sampling

CONTACTS AND LOCATIONS:
Overall Officials: Ove J Nielsen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, Hematology clinic, Copenhagen
  - Herlev Hospital, Hematology Clinic, Herlev